CLINICAL TRIAL: NCT05144126
Title: Safety, Radiological and Patient Reported Outcomes of i-FACTOR+ Matrix Bone Graft Device - A Canadian, Multicenter, Post-Market Clinical Investigation
Acronym: CAPREG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CeraPedics, Inc (Industry)
Collaborators: Talosix (Unknown); Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21/SP/COM/01
Record Dates: First submitted 2021-11-21; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- i-Factor Arm (Experimental): All patients undergoing spine fusion surgery will be treated with i-FACTOR
  Interventions: Other: CT radioraphic assessment

INTERVENTIONS:
Other: CT radioraphic assessment — CT radioraphic assessment

SUMMARY:
The study intends tracking the usage patterns of a Bonegraft device within spine surgery in a multicenter setting in Canada.

DETAILED DESCRIPTION:
The study wil track the usage patterns of a bone graft by identifying and classifying spine surgery procedures by access and segment type within the spins and furthet, record and analyse safety and performance measures associated with each classification. This is a post-market surveillance study

ELIGIBILITY:
Inclusion Criteria:

* Adult patient subjects not responding to conservative management of neck / arm or back/leg pain and requiring spinal fusion between levels C1 - T2 or L1 - S1
* Informed Consent

Exclusion Criteria:

* Hypersensitivity to i-FACTOR Bone Graft Devices
* Adult Spinal deformity, Spinal Cord Injury
* Infection
* Compromised renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
index segment revision | 12-months post-operative
  Reintervention rate at index segment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Witiw, MD, Principal Investigator — St Michael's Hosptal Toronto

IPD SHARING:
Plan to Share IPD: No